CLINICAL TRIAL: NCT03768921
Title: Use of Electrical Impedance Tomography in Children With Syndrome of Acute Respiratory Disorder
Brief Title: Ventilatory Monitoring in Children With Respiratory Distress Syndrome With Electrical Impedance Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Department of Movement Human Sciences Coordinator, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 78745217.8.0000.5171
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: Dyspnea; Respiration, Artificial; Intensive Care Units
MeSH Terms: conditions — Respiratory Distress Syndrome; Dyspnea; Respiratory Aspiration

STUDY DESIGN:
Masking Description: The research design is a longitudinal, quantitative and analytical clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP Titriation (Experimental): patients with respiratory distress syndrome will undergo alveolar recruitment in the mechanical ventilator and will have their final positive mechanical ventilator pressure determined by ventilator evaluation by the electrical impedance tomograph. The increase of the peep in the mechanical ventilator to perform the alveolar recruitment will be of 2 in 2 cmH2O every 2 minutes until the pressure reaches 25 cmH20, after the pressure was reduced in the same way being evaluated in the tomograph what will be the point with greater alveolar recruitment, having greater ventilation, without alveolar hyperdistension or alveolar collapse.
  Interventions: Other: PEEP Titriation

INTERVENTIONS:
Other: PEEP Titriation — The alveolar recruitment maneuver PEEP reaches a maximum of 25 cmH2O, with recruitment being performed progressively, where the pressure variation is maintained at 15 cmH2O and the PEEP increase progressively occurs at 2 cmH2O every 2 minutes and Ventilatory mode with Controlled Pressure Ventilation. After the alveolar recruitment maneuver, the PEEP titration or determination will be performed, where the PEEP of 2 cmH2O will be reduced every 2 minutes and the variables after the alveolar recruitment maneuver and PEEP maintenance will be checked in the TIMPEL brand equipment at the point where the patient has better alveolar recruitment, with fewer alveolar collapsing points and pulmonary hyperdistension.

SUMMARY:
INTRODUCTION: Electrical impedance tomography is a tool for noninvasive monitoring of pulmonary ventilation in real time, which is used during alveolar recruitment maneuvers in patients with acute respiratory distress syndrome. OBJECTIVES: To identify ventilatory and hemodynamic changes during the alveolar recruitment maneuver in children with acute respiratory distress syndrome using electrical impedance tomography. METHODS: Twenty children, aged 4 to 12 years, who present a diagnosis of respiratory distress syndrome, with indication of alveolar recruitment admitted to the Pediatric Intensive Care Unit of the Santa Casa de Misericórdia Foundation of Pará will be selected. Data collection will consist of three before the alveolar recruitment maneuver, immediately after the alveolar recruitment maneuver, 2 hours after the alveolar recruitment maneuver, where the pulmonary ventilation distribution, the driving pressure, the real-time reading compliance will be analyzed. tomography of the Timpel brand, autonomic heart rate modulation through the Polar® RS800CX device, physiological variables such as heart rate, oxygen pulse saturation and blood pressure by measuring the DIXTAL multi-parameter monitor, blood oxygen pressure and the oxygen content dog. The statistical analysis will be performed in the Biostat 5.2 program, and the choice of tests will depend on the types of distributions found and the homogeneity of the respective variances.

DETAILED DESCRIPTION:
The present study will be developed at the referral hospital in the north of the country, Santa Casa de Misericórdia Foundation of Pará, located at Rua Bernal do Couto 992, Bairro Umarizal, Belém (PA), Unit of Intensive Pediatric Therapy, with the participation of the unit's interdisciplinary team. The data collection period will take place between December 2017 and February 2019.

For the measurement of ventilatory variables (static and regional compliance, regional ventilation, driving pressure, alveolar hyperdistension, alveolar collapse and PEEP titration), the Timpel® Brand Electrical Impedance Tomography monitor will be used to measure hemodynamic variables arterial and oxygen pulse saturation) a DIXTAL® brand monitor will be used.

The instruments used to measure HRV will be the Polar® RS800CX device that features WearLink heart rate sensor, elastic band, contact gel, interface with USB input and a computer.

After the selection and acceptance of the terms of consent and clarification of doubts the research will be carried out in four stages, where the first one will start before performing the alveolar recruitment maneuver; the second, during the alveolar recruitment maneuver; the third, 24 hours after the alveolar recruitment maneuver; and the fourth 48 hours after the alveolar recruitment maneuver. Each of said steps will be divided into sub-steps according to the procedures.

Before the beginning of the alveolar recruitment maneuver, the minor will be sedated and curarized, in order to avoid interference in the recruitment protocol and thus increase the incidence of complications such as increased intrathoracic pressure and consequent alveolar rupture.

Next, the ventilator mechanic flow sensor will be coupled between the child's orotracheal tube that is intubated and the reference sensor on the right flank of the patient's abdomen. The Electrical Impedance Tomography will be connected and observed if all the electrodes are coupled to the patient's chest. At this moment the hemodynamic and ventilatory variables of the study will be collected.

The alveolar recruitment maneuver based on the study of Borges et al. (2006), modified so that PEEP reaches a maximum of 25 cmH2O, with recruitment being performed progressively, as demonstrated in Figure 2, where the pressure variation is maintained at 15 cmH2O and the PEEP increase progressively occurs at 2 cmH2O every 2 minutes, with respiratory rate set at 15 breaths per minute and Ventilatory mode with Controlled Pressure Ventilation ( PCV). After the alveolar recruitment maneuver, the PEEP titration or determination will be performed, where the PEEP of 2 cmH2O will be reduced every 2 minutes and the variables after the alveolar recruitment maneuver and PEEP maintenance will be checked in the TIMPEL brand equipment at the point where the patient has better alveolar recruitment, with fewer alveolar collapsing points and pulmonary hyperdistension. This PEEP is maintained for 24 hours so that alveolar recruitment is not lost. The variables will be evaluated again in 24 hours and 48 hours after the alveolar recruitment maneuver to identify the benefits of the same.

For the collection of the modulation will be performed the analysis of the HRV where initially the electrodes of the elastic strip will be moistened with contact gel, then the WearLink sensor will be connected to the band that will be positioned around the patient's chest, just below the pectoral muscles and the hook will be attached to the other end of the strip, subsequently the length of the strip will be adjusted so that the strip is juxtaposed to the skin, yet comfortable. It will be checked if the wetted areas of the electrodes are in contact with the skin and if the Polar logo on the connector is centered and straight. The volunteer will then be placed in the supine position, his / her Systemic Arterial Pressure (BP) will be measured, and then the patient will be advised not to talk, sleep, move his arms or cough during the test.

Once the above procedures have been completed, the R-R intervals will be captured, which will last 10 minutes, where the FR will be marked every minute. At the end, BP will be measured again in the supine position. Then the RS800CX interface will be placed in the computer's USB port and the sensor will be placed next to it for infrared data capture. In this way the data will be downloaded and stored with the patient's name and the day of collection in the Softwere Polar ProTreiner 5. Then the data will be transformed into .txt format and submitted to the Kubios HRV 2.2 softwere software to analyze the heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS, aged 7 to 12 years;
* Indication of treatment with alveolar recruitment maneuver.

Exclusion Criteria:

* Clinical condition that does not allow alveolar recruitment maneuvers
* Severe hypotension
* Cardiac arrhythmia
* Pneumothorax
* Pneumatocele untreated.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Driving pressure | evaluation during two days
  The driving pressure, which indicates alveolar pressure variation and alveolar distension capacity, will be evaluated.
Alveolar collapse | evaluation during two days
  the percentage of alveolar collapse, which indicates how much the pulmonary alveolus is without air.
Alveolar hiperdistension | Evaluation during two days
  the percentage of hyperdistended alveoli, which indicates that the alveoli are with excess air in their interior.
Regional air ventilation | Evaluation during two days
  Regional air ventilation, which indicates how air is distributed in the lung, demonstrating the most ventilated and least ventilated areas in the lung.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Rocha, Phd, Principal Investigator — Universidade do Estado do Pará
Locations (1):
- Fundação Santa Casa de Misericórdia do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hamm LF, Wenger NK, Arena R, Forman DE, Lavie CJ, Miller TD, Thomas RJ. Cardiac rehabilitation and cardiovascular disability: role in assessment and improving functional capacity: a position statement from the American Association of Cardiovascular and Pulmonary Rehabilitation. J Cardiopulm Rehabil Prev. 2013 Jan-Feb;33(1):1-11. doi: 10.1097/HCR.0b013e31827aad9e. PMID 23254246
- [Result] Yehya N, Thomas NJ. Disassociating Lung Mechanics and Oxygenation in Pediatric Acute Respiratory Distress Syndrome. Crit Care Med. 2017 Jul;45(7):1232-1239. doi: 10.1097/CCM.0000000000002406. PMID 28350644
- [Result] Ward SL, Quinn CM, Valentine SL, Sapru A, Curley MA, Willson DF, Liu KD, Matthay MA, Flori HR. Poor Adherence to Lung-Protective Mechanical Ventilation in Pediatric Acute Respiratory Distress Syndrome. Pediatr Crit Care Med. 2016 Oct;17(10):917-923. doi: 10.1097/PCC.0000000000000903. PMID 27513687
- [Result] Kheir JN, Walsh BK, Smallwood CD, Rettig JS, Thompson JE, Gomez-Laberge C, Wolf GK, Arnold JH. Comparison of 2 lung recruitment strategies in children with acute lung injury. Respir Care. 2013 Aug;58(8):1280-90. doi: 10.4187/respcare.01808. Epub 2012 Dec 4. PMID 23232733
- [Result] Donoso F A, Arriagada S D, Diaz R F, Cruces R P. [Ventilation strategies in the child with severe hypoxemic respiratory failure]. Gac Med Mex. 2015 Jan-Feb;151(1):75-84. Spanish. PMID 25739487